CLINICAL TRIAL: NCT03705832
Title: Ginger's Therapeutic Potential in Asthma
Acronym: GINGER
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emily DiMango, MD (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Emily DiMango, MD, Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAR8427; R61AT009989 (NIH)
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Asthma
Keywords: Ginger; Dietary supplement
MeSH Terms: conditions — Asthma | interventions — ginger extract

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active drug (Experimental): Subjects assigned to the intervention will receive 2 grams daily of Ginger Extract for 56 days.
  Interventions: Drug: Ginger Extract
- Placebo (Placebo Comparator): Subjects assigned to the placebo group will receive a matching placebo for 56 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginger Extract — 2gm Capsule of Ginger extract
  Other Names: Ginger
  Arms: Active drug
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo controlled study to study whether there are potential benefits of consuming ginger by individuals with asthma.

DETAILED DESCRIPTION:
Presently an estimated 25.9 million Americans suffer from asthma and over half have at least one asthma attack per year. Recent studies found that 60% of moderate asthmatics and 70% of severe asthmatics report using complementary and alternative medicine (CAM) to self-treat their asthma symptoms.The exact mechanism of action of these agents is unclear but may involve attenuation of allergic response, anti-inflammatory and antioxidant effects, and/or direct effects on airway smooth muscle which are responsible for airway narrowing in asthma.

Studies done in mouse models of asthma and directly on airway smooth muscle cells demonstrate that ginger blocks one of the critical inflammatory pathways in asthma and thus leads to reduced airway inflammation and relaxation of airway smooth muscle. Clinical trials with chronic oral ginger therapy in humans have demonstrated safe consumption of 2 grams per day for 28 days with demonstrated anti-inflammatory effects in colon cancer and inflammatory bowel diseases. Thus, the investigators hypothesize that oral ginger at a dose of 2 grams per day will reduce airway inflammation and will reduce serum levels of asthma related inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women age 18 or older;
2. Treatment with inhaled corticosteroids (ICS) +/- long acting β-agonists/long acting muscarinics and montelukast;
3. Physician diagnosed asthma;
4. Forced expiratory volume (FEV1) ≥60% of predicted
5. Methacholine PC(20) < 16 mg/ml if taking ICS and < 8mg/ml if not taking ICS at Visit 2.
6. Non-smoker (e.g., tobacco, e-cigarette, marijuana) for ≥1 yr.;
7. ≤10 pack-year smoking history;
8. Suboptimal control of asthma as determined by a score < 19 or less on the Asthma Control Test (ACT) at Screening Visit (Visit 1) and Randomization Visit (Visit 3).

Exclusion Criteria:

1. Other major chronic illnesses: Conditions which in the judgment of the study physician would interfere with participation in the study, e.g., non-skin cancer, uncontrolled diabetes mellitus, coronary artery disease, congestive heart failure, stroke, severe hypertension, renal failure, liver disorders, malabsorption disorders, immunodeficiency states, major neuropsychiatric disorder;
2. Cardiovascular problems: Myocardial infarction or stroke in last 3 months Uncontrolled hypertension Known aortic aneurysm
3. History of physician diagnosis of chronic bronchitis, emphysema or chronic obstructive pulmonary disease (COPD)
4. Medication use: Current consumption of ginger supplements, oral corticosteroid use within the past 6 weeks, use of an investigational treatment in the previous 30 days, known adverse reaction to ginger or ginger products;
5. Females of childbearing potential: Pregnant or lactating; participants of appropriate age who might be pregnant at the time of enrollment will be screened with urine pregnancy tests at each visit and cannot participate if pregnant. Participants must agree to use effective contraception during the trial.
6. Inability to perform acceptable and repeatable spirometry maneuvers throughout the test procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily DiMango, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Asthma Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 54 participants were enrolled and 12 participants were excluded due to: lost to follow-up, asthma controlled, lung function below threshold, on exclusionary medications, and not taking asthma medications. Eight participants were withdrawn due to an institutional COVID-19 research pause.
Period: Overall Study
Arm/Group | Active Drug | Placebo
Started | 21 | 13
Completed | 20 | 12
Not Completed | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug | Placebo | Total
Number analyzed (Participants) | 20 | 12 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (17.5) | 56.1 (13) | 54.7 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 9 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 9 | 3 | 12
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Tolerance to Inhaled Methacholine
Description: A methacholine challenge test is a medical test used to assist in the diagnosis of asthma. The patient breathes in nebulized methacholine at gradually increasing doubling doses, starting with diluent only. Methacholine provokes bronchoconstriction, or narrowing of the airways via M3 receptors. The degree of narrowing can then be quantified by spirometry which is performed after inhalation of each dose. Methacholine provocation dose (PD)20 values will be used to measure any change in airway hyperresponsiveness.
Time Frame: Baseline and Day 28
Population: Nine active drug and seven placebo participants were analyzed due to: 1) low lung function at the time of the study visit (methacholine testing was withheld for safety reasons) and 2) during the COVID-19 pandemic, methacholine testing was discontinued, as it is an aerosol generating procedure.
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 9 | 7
mg/ml | 5.3 (15.1) | 24.2 (55.9)

2. Primary Outcome: Change in Tolerance to Inhaled Methacholine
Description: A methacholine challenge test is a medical test used to assist in the diagnosis of asthma. The patient breathes in nebulized methacholine at gradually increasing doubling doses, starting with diluent only. Methacholine provokes bronchoconstriction, or narrowing of the airways via M3 receptors. The degree of narrowing can then be quantified by spirometry which is performed after inhalation of each dose. Methacholine provocation dose (PD20) values will be used to measure any change in airway hyperresponsiveness.
Time Frame: Baseline and Day 56
Population: Twelve active drug and three placebo participants were analyzed due to: 1) low lung function at the time of the study visit (methacholine testing was withheld for safety reasons) and 2) during the COVID-19 pandemic, methacholine testing was discontinued, as it is an aerosol generating procedure.
Measure: Mean (Standard Deviation); unit: PD20 of methacholine (mg/ml)
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 12 | 3
PD20 of methacholine (mg/ml) | 4 (13.1) | 78.4 (137.9)

3. Primary Outcome: Change in Fractional Exhaled Nitric Oxide (FeNO)
Description: Measure of markers of asthmatic lung inflammation
Time Frame: Baseline and Day 28
Population: Eight placebo analyzed due to device malfunction.
Measure: Mean (Standard Deviation); unit: fractional exhaled parts per billion
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 20 | 8
fractional exhaled parts per billion | 8.5 (26.9) | 20.1 (43.1)

4. Primary Outcome: Change in Fractional Exhaled Nitric Oxide (FeNO)
Description: Measure of markers of asthmatic lung inflammation
Time Frame: Baseline and Day 56
Population: Nine placebo analyzed due to device malfunction.
Measure: Mean (Standard Deviation); unit: fractional exhaled parts per billion
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 20 | 9
fractional exhaled parts per billion | -4.6 (20.4) | 26.2 (62.6)

5. Secondary Outcome: Change in Serum Cytokines
Description: Measure of markers of asthmatic lung inflammation
Time Frame: Baseline and Day 56
Population: Cytokine samples were collected from 15 and 10 active and placebo participants respectively.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 15 | 10
pg/ml | -1.297 (18.81) | 2.411 (18.81)

6. Secondary Outcome: Change in Eosinophilia
Description: Measure of markers of asthmatic lung inflammation
Time Frame: Baseline and Day 56
Measure: Mean (Standard Deviation); unit: x10^9 cells/L
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 20 | 12
x10^9 cells/L | 0.007 (0.219) | 0.128 (0.211)

7. Secondary Outcome: Change in Score on the Asthma Control Test (ACT)
Description: Asthma symptom score will be measured with the Asthma Control Test at Visit 1, 2 and 5.This instrument, which has been validated for ages 12-84 years, is a 4-week recall questionnaire that addresses issues of asthma control, symptoms, and nocturnal awakenings. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Time Frame: Baseline and Day 56
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 20 | 12
score on a scale | -1.6 (3.966) | -2.0 (2.045)

8. Secondary Outcome: Change In Score on Juniper Mini-Asthma Specific Quality of Life (Mini AQLQ-J)
Description: This questionnaire consists of 15 items in 4 domains with a 2-week recall period. Scores range from 7-105, with higher scores indicating better quality of life.
Time Frame: Baseline and Day 56
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 20 | 12
score on a scale | -11.3 (21.91) | -11.5 (13.01)

ADVERSE EVENTS:
Time Frame: Up to Day 78
Arm/Group | Active Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/12
Other Adverse Events (participants affected / at risk) | 0/20 | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Drug (N=20) | Placebo (N=12)
Coronavirus Disease 2019 (COVID-19) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Drug (N=20) | Placebo (N=12)
Absence Seizure (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03705832/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT03705832/ICF_000.pdf